CLINICAL TRIAL: NCT05622643
Title: Very High Definition Cohort: Assessment of New Prognostic Biomarkers of Disability Worsening in a Multicenter Cohort of MS Patients by Imaging, Optical Coherence Tomography and Biology
Brief Title: OFSEP Very High Definition Cohort
Acronym: VHD cohort
Status: Recruiting | Type: Observational
Sponsor: EDMUS Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 004
Record Dates: First submitted 2022-10-11; First posted 2022-11-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: Prognostic factors; MS progression; MRI; OCT; NFL; GFAP
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MS: 250 patients with MRI, OCT and bio sample
  Interventions: Other: MRI
- Healthy subjects: 50 healthy subjects with MRI
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Comparison between groups

SUMMARY:
Multiple sclerosis (MS) is the most common acquired neurological disease leading to disability in young adults. MS often leads to the development of a physical and/or cognitive impairment that disables patients in their daily lives. Early use of disease modifying treatments for patients at risk of developing disability is therefore essential.

However, disability progression is very heterogeneous between patients and currently impossible to predict at the individual level. Thus, numerous studies, particularly epidemiological and imaging studies, have identified prognostic factors for the development of disability such as age, gender, number of relapses during the first years of the disease, existence of a residual disability after a first relapse, number of gadolinium-enhancing lesions on initial MRI, early brainstem and spinal cord lesions. However, these different factors only explain incompletely the progression of the physical or cognitive disability in MS patients. In particular, some components of MS pathophysiology, more related to the progressive development of disability, such as axonal degeneration or the existence of chronic inflammation of the central nervous system (CNS) are usually not measured by these biomarkers.

In this research project, the investigators will test promising biomarkers, focused on these components of the disease, on a large cohort of patients in a multicenter setting, in order to evaluate their added value to predict disability progression, in comparison with more classical biomarkers such as clinical characteristics, and brain and spinal cord lesion load.

In particular, the investigators will test:

* Imaging biomarkers extracted from brain and spinal cord MP2RAGE, brain and spinal cord QSM, brain and spinal cord relaxometry, brain diffusion and spinal cord magnetization transfer sequences
* Biomarkers extracted from optical coherence tomography (OCT)
* Biological biomarkers (serum neurofilament-light chain (NFL) and Glial Fibrillary Acidic Protein (GFAP))

ELIGIBILITY:
For MS patients:

* Inclusion Criteria:

  * The patient must be already included in the OFSEP High Definition cohort (NCT03603457).
  * The patient must have given his informed and signed consent for the inclusion in the VHD cohort.
  * The patient must be insured or beneficiary of a health insurance plan.
* Exclusion Criteria:

  * The patient is under judicial protection.
  * The patient refuses to sign the consent.
  * It is impossible to correctly inform the patient (Inability to understand the study, language problem).
  * The patient has experienced a relapse in the previous 3 months.
  * The patient is pregnant or breast-feeding (MRI contraindicated).
  * Patient with MRI contra-indications (patient with a pacemaker, ferromagnetic vascular clip, infusion pump, neurostimulator, cochlear implants or in whom there is a suspicion of a metallic foreign body).
  * The patient has a severe psychiatric illness
  * The patient has severe chronic alcoholism

For healthy subjects:

* Inclusion Criteria:

  * The healthy subject must be older than 18 years
  * The healthy subject must have given his informed and signed consent for the inclusion in the VHD cohort.
  * The healthy subject must be insured or beneficiary of a health insurance plan.
* Exclusion Criteria:

  * The healthy subject is under judicial protection.
  * It is impossible to correctly inform the healthy subject (Inability to understand the study, language problem).
  * The healthy subject is pregnant or breast-feeding (MRI contraindicated).
  * The healthy subject has MRI contra-indications (a pacemaker, ferromagnetic vascular clip, infusion pump, neurostimulator, cochlear implants or in whom there is a suspicion of a metallic foreign body).
  * The healthy subject has a history of disease that may affect the central nervous system.
  * The healthy subject has a family history of MS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In order to ensure the inclusion of patients with different MS phenotypes representative of the general MS patients population in the VHD cohort, the investigators will aim to respect the inclusion percentages of at least 10% of patients with primary progressive MS and at least 15% of patients with secondary progressive MS.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Global disability progression | 2 years
  Global disability progression will be scored by the Expanded disability score system (EDSS). Disability progression will be defined as an increase in the EDSS of at least 1 point if the baseline EDSS was 5.5 or less, or 0.5 point if the Baseline EDSS was

SECONDARY OUTCOMES:
Composite disability progression score | 2 years
  A composite disability progression score will be defined as an increase in the EDSS score, or an increase in the time to perform the timed 25-foot walk ≥ 20%, or an increase in the time to complete the 9-hole peg test ≥ 20% at 2 years compared to baseline
Change in the Symbol Digit Modalities Test score | 2 years
  Change in the Symbol Digit Modalities Test (SDMT) score from baseline to 2-year
Change in the American Spinal Cord Injury Association motor sub-score | 2 years
  Change in the American Spinal Cord Injury Association (ASIA) motor sub-score from baseline to 2-year
Focal inflammatory activity | 2 years
  Focal inflammatory activity at 2 years will be defined by the occurrence of a clinical relapse and/or MRI activity (new T2 lesion)
No evidence of disease activity 3 | 2 years
  No evidence of disease activity (NEDA) 3 at 2 years will be defined as no evidence of disability progression scored by the EDSS, relapse, MRI activity
Between-subject, between-center and between-session coefficient of variation of measurements extracted quantitative MRI | At inclusion
  Between-subject, between-center and between-session coefficient of variation (in percentage) of measurements extracted from baseline brain and spinal cord quantitative MRI (T1, Myelin water fraction, magnetization transfer ratio, parameters extracted from diffusion imaging)
Number of brain and spinal cord lesion detected using 3D MP2RAGE sequence and the classical OFSEP sequences at baseline and 2 year | At inclusion and 2 years
Number of new brain and spinal cord lesion detected at 2 years using 3DMP2RAGE sequence and the classical OFSEP sequences | 2 years
Number of detected brain and spinal cord lesions per patient and per expert with and without the automatic tool at baseline and 2 year | At baseline and 2 year

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU de Lyon, Lyon
  - CHU de Nancy, Nancy
  - CHU de Nîmes, Nîmes
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
URL: http://www.ofsep.org/en/data-access